CLINICAL TRIAL: NCT07244159
Title: Effects of Dynamic Surface Exercise Training on Functional Mobility, Balance and Coordination in Children With Diplegic Cerebral Palsy
Brief Title: Effects of Dynamic Surface Exercise Training in Children With Diplegic Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/HAFIZA IRAM BATOOL
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Child, Only
Keywords: Diplegic cerebral palsy; Dynamic surface exercise training; Balance; Coordination; Gross Motor Function Measure (GMFM)
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: This is a randomized clinical trial,total of 14 children with diplegic cerebral palsy of age between 6 and 8 years of both genders with Gross Motor Function Classification System of level III and IV will be recruited to participate in randomized controlled study. The study will be completed within 10 months after the approval of the synopsis. Technique of the study is non-probability convenient sampling technique. Recruited will be randomly divided into two groups, dynamic surface exercise training (DSET) group and standard physiotherapy training group. Both the groups receive active training program lasting for 60 minutes, 4 days/week for 6 weeks who have the ability to follow and accept verbal instructions. Gross Motor Function Measure (GMFM)-88 and Pediatric Balance Scale (PBS) and Time up and go test scores will be recorded at baseline, and at the end of 6-week post-intervention.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols efforts will be put to mask the both groups about the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): This group will be given dynamic surface exercise training lasting for 60 minutes, 4 days /week for 6 weeks. For balance, the first (simple) level included supine abdominal draw-in (20 repetitions), abdominal draw-in with both knees to the chest (10e20 repetitions), and supine twist (10e20 repetitions) . The second (medium) level included pelvic bridging (3e5 repetitions) and twist with a medicine ball (10e20 repetitions)
  Interventions: Other: Dynamic surface exercise training
- Group B (Active Comparator): This group will be given standard physiotherapy training lasting for 60 minute, 4 days/week for 6 weeks. Standard physiotherapy includes side sitting on bench/stool to quadruped-quadruped to side sit (transition activity) 5 times each side and 1 set in a day. On bench, patient forward bend and pick the ball, come back to sitting and through the ball for 10 times and 1 set
  Interventions: Other: Standard physiotherapy Training

INTERVENTIONS:
Other: Dynamic surface exercise training — This group will be given dynamic surface exercise training lasting for 60 minutes, 4 days /week for 6 weeks. For balance, the first (simple) level included supine abdominal draw-in (20 repetitions), abdominal draw-in with both knees to the chest (10e20 repetitions), and supine twist (10e20 repetitions) . The second (medium) level included pelvic bridging (3e5 repetitions) and twist with a medicine ball (10e20 repetitions). Finally, the third (difficult) level included bridging with the head on a physio ball (the position was held for 3e5 s, followed by a slow relaxation phase, with 10e20 repetitions) and prone bridging (the entire sequence was repeated 3e5 times.
  Arms: Group A
Other: Standard physiotherapy Training — This group will be given standard physiotherapy training lasting for 60 minute, 4 days/week for 6 weeks. Standard physiotherapy includes side sitting on bench/stool to quadruped-quadruped to side sit (transition activity) 5 times each side and 1 set in a day.
  Arms: Group B

SUMMARY:
Data will be collected after the approval of synopsis a total of 14 children with diplegic cerebral palsy of age between 6 and 8 years of both genders with Gross Motor Function Classification System of level III and IV will be recruited to participate in randomized controlled study. The study will be completed within 10 months after the approval of the synopsis. Technique of the study is non-probability convenient sampling technique. Recruited will be randomly divided into two groups, dynamic surface exercise training (DSET) group and standard physiotherapy training group. Both the groups receive active training program lasting for 60 minutes, 4 days/week for 6 weeks who have the ability to follow and accept verbal instructions. Gross Motor Function Measure (GMFM)-88 and Pediatric Balance Scale (PBS) and Time up and go test scores will be recorded at baseline, and at the end of 6-week post-intervention.

DETAILED DESCRIPTION:
This group will be given dynamic surface exercise training lasting for 60 minutes, 4 days /week for 6 weeks. For balance, the first (simple) level included supine abdominal draw-in (20 repetitions), abdominal draw-in with both knees to the chest (10e20 repetitions), and supine twist (10e20 repetitions) . The second (medium) level included pelvic bridging (3e5 repetitions) and twist with a medicine ball (10e20 repetitions). Finally, the third (difficult) level included bridging with the head on a physio ball (the position was held for 3e5 s, followed by a slow relaxation phase, with 10e20 repetitions) and prone bridging (the entire sequence was repeated 3e5 times).

This group will be given standard physiotherapy training lasting for 60 minute, 4 days/week for 6 weeks. Standard physiotherapy includes side sitting on bench/stool to quadruped-quadruped to side sit (transition activity) 5 times each side and 1 set in a day. On bench, patient forward bend and pick the ball, come back to sitting and through the ball for 10 times and 1 set. On floor, standing: throwing and catching the ball from different direction, 10 times each side, 1 set Gross motor function measure-88 and pediatric balance scale and time up and go test scores will be recorded at baseline, and at the end of 6-week post-intervention

ELIGIBILITY:
Inclusion Criteria:

* Age between 5 and 8 years of both genders
* Classification as level III and IV on the Gross Motor Function Classification system (GMFCS)

Exclusion Criteria:

* • Any orthopedic surgery or botulinum toxin injection in the past 6 months.

  * Refusal by the parents to participate.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measure (GMFM) | baseline, 1st week and 6th week
  Balance Scale (PBS) will be the outcome measures use in this trial. GMFM-88 has excellent relative reliability of excellent (Intraclass correlation coefficient (ICC) = 0.952-1.000)
Pediatric Berg Balance Scale | baseline, 1st week and 6th week
  The Pediatric Balance Scale is a modified version of the Berg Balance Scale that is used to assess functional balance skills in school-aged children
Time up and go test | baseline, 1st week and 6th week
  Reliability of TUG test was high, with ICC of 0.99 for within-session reliability and 0.99 for test-retest reliability

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Iram Batool, MS-PT, Principal Investigator — Riphah International University
Locations (1):
- Hafiza Iram Batool, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salphale VG, Kovela RK, Qureshi MI, Harjpal P. Effectiveness of Pelvic Proprioceptive Neuromuscular Facilitation on Balance and Gait Parameters in Children With Spastic Diplegia. Cureus. 2022 Oct 22;14(10):e30571. doi: 10.7759/cureus.30571. eCollection 2022 Oct. PMID 36415346